CLINICAL TRIAL: NCT04665180
Title: Determinants for Return to Work After Primary Knee Arthroplasty: a Prospective Study
Brief Title: Determinants for Return to Work After Primary Knee Arthroplasty
Acronym: RTW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S63495
Record Dates: First submitted 2020-12-01; First posted 2020-12-11 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-09

CONDITIONS: Knee Arthropathy; Return to Work

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary knee arthroplasty (Experimental): Questionnaires
  Interventions: Diagnostic Test: Primary knee arthroplasty

INTERVENTIONS:
Diagnostic Test: Primary knee arthroplasty — Patients who return to work after primary knee arthroplasty

SUMMARY:
The increase of end-stage osteoarthritis (OA) in an increasingly younger population is directly correlated with the rising incidence of obesity. As a result, knee arthroplasty (KA), which is a definitive end-stage treatment option, is increasingly performed on working age people. Knowledge and understanding of the underlying factors that drive the ability for people to return to work is crucial.

First and foremost, the investigators would have like to have a clear idea of the percentage of patients who return to work and at what time postoperatively. The investigators would also determine the different factors influencing employment in the patient population after undergoing a knee arthroplasty and register the evolution in the necessity of pain medication pre-and postoperatively. Ideally, the investigators can include a short questionnaire regarding return to sports to gather valuable information.

DETAILED DESCRIPTION:
The increase of end-stage osteoarthritis (OA) in an increasingly younger population is directly correlated with the rising incidence of obesity. As a result, knee arthroplasty (KA), which is a definitive end-stage treatment option, is increasingly performed on working age people. Knowledge and understanding of the underlying factors that drive the ability for people to return to work is crucial.

First and foremost, the investigators would have like to have a clear idea of the percentage of patients who return to work and at what time postoperatively. The investigators would also determine the different factors influencing employment in the patient population after undergoing a knee arthroplasty and register the evolution in the necessity of pain medication pre-and postoperatively. Ideally, the investigators can include a short questionnaire regarding return to sports to gather valuable information.

Adult patients with an indication for primary knee arthroplasty (total + unicondylar) can take part in the study. This will be decided by clinical examination and radiographic evaluation, having the result of the previous therapies and the patient-specific needs in mind (standard of care). The patients have to be younger than or equal to 63 years old at the time of surgery and actively been working 2 years prior to surgery.

In line with the standard of care, the patients will be seen after 4-8 weeks, 3-4 months and 1 year postoperatively. Radiological examinations are foreseen at 4-8 weeks and 1 year postoperatively (standard of care). Pre-operatively, a general questionnaire is filled in by the patients. The patient questionnaires Knee Society Score (KSS), Knee Injury and Osteoarthritis Outcome Score (KOOS), Forgotten Knee Joint Score, Quickscan, Work, Osteoarthritis and joint-Replacement Questionnaire (WORQ) will be filled in by the patients during the screening visit and on each consultation at 4-8 weeks, 3-4 months, 6 months, 1 year and 1,5 year. The Tegner score will be filled in by the patients pre-operatively and at 1 year postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Primary knee arthroplasty (total + unicondylar)
* Patients younger than or equal to 63 years old at the time of surgery
* Actively been working 2 year prior to surgery.

Exclusion Criteria:

* No informed consent
* Revision surgery
* Patients older than 63 years of age at the time of surgery
* Patients who haven't were unable to work due to other, non-knee related, health issues

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Quickscan questionnaire | Time frame of 1,5 year postoperatively
  Return to work is measured using the Quickscan questionnaire during screening visit, at 4-8 weeks, 3-4 months, 6 months, 1 year and 1,5 year.
  In the Quickscan questionnaire, all questions are scored ranging from "0" totally disagree to "5" totally agree.
Work, Osteoarthritis and joint-Replacement Questionnaire (WORQ) | Time frame of 1,5 year postoperatively
  Return to work is measured using the Work, Osteoarthritis and joint-Replacement Questionnaire (WORQ) during screening visit, at 4-8 weeks, 3-4 months, 6 months, 1 year and 1,5 year.
  The WORQ is a patient reported outcome measure (PROM) in which the patient indicates his experiences in 13 knee-stressing activities in the past week by scoring the difficulty the patient experienced. A formula is used to calculate the total score that ranges from 0 ('very much difficulty/ can't do') to 4 ('no difficulty at all').

SECONDARY OUTCOMES:
Knee rate and patient's functional abilities | within a time frame of 1,5 year postoperatively
  To rate the knee and patient's functional abilities, the Knee Society Score (KSS) is used during screening visit, at 4-8 weeks, 3-4 months, 6 months, 1 year and 1,5 year.
Knee symptoms | within a time frame of 1,5 year postoperatively
  Knee symptoms are measured using Knee Injury and Osteoarthritis Outcome Score (KOOS) during screening visit, at 4-8 weeks, 3-4 months, 6 months, 1 year and 1,5 year.
Awareness of knee joint/knee prothesis in daily life | within a time frame of 1,5 year postoperatively
  Be aware of knee joint/knee prothesis in daily life is measured using the Forgotten Knee Joint Score during screening visit, at 4-8 weeks, 3-4 months, 6 months, 1 year and 1,5 year.
Return to sports | within a time frame of 1 year postoperatively
  Return to sports is measured using the Tegner score during screening visit and at 1 year postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Hilde Vandenneucker, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No